CLINICAL TRIAL: NCT05274620
Title: Integrating a Suite of Mental Health Apps for Depression in a Healthcare Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adaptive Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R44MH114725-05 (NIH)
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IntelliCare (Other): 8 weeks of IntelliCare
  Interventions: Behavioral: IntelliCare

INTERVENTIONS:
Behavioral: IntelliCare — A mobile intervention that use principles of computerized therapy to decrease symptoms of depression

SUMMARY:
The purpose of this study is to evaluate the implementation of IntelliCare as a frontline intervention within health care settings.

DETAILED DESCRIPTION:
This study will evaluate the implementation of IntelliCare in two settings: Primary care in the McLeod Health system, serving a rural population where mental healthcare workers are scarce, and Northwestern Medicine's Department of Psychiatry, which currently has a 9-month waitlist for psychological services.

ELIGIBILITY:
Inclusion Criteria:

* Patient who have been identified as depressed or anxious by a care provider in one of the participating healthcare organizations.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Reach | 5 months
  1. Number of eligible patients during trial period; 2) number offered IntelliCare; 3) number initiating IntelliCare; 4) number completing IntelliCare
Cost | 7 months
  Cost of delivering IntelliCare per patient

SECONDARY OUTCOMES:
Depression | Administered weekly over 8 weeks
  Patient Health Questionnaire-9 (PHQ-9); higher scores indicate greater symptom severity

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn MacIver, Principal Investigator — Adaptive Health, Inc
Locations (2):
- United States (2):
  - Northwestern Medicine Dept of Psychiatry, Chicago, Illinois
  - MacLeod HealthCare, Florence, South Carolina

IPD SHARING:
Plan to Share IPD: No